CLINICAL TRIAL: NCT04322708
Title: A Phase 2/3, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Lirentelimab (AK002) in Adult and Adolescent Patients With Active Eosinophilic Esophagitis
Brief Title: A Study of Lirentelimab (AK002) in Patients With Active Eosinophilic Esophagitis
Acronym: KRYPTOS
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Allakos Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AK002-014
Record Dates: First submitted 2020-03-24; First posted 2020-03-26 (Actual); Results first posted 2024-01-02 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Eosinophilic Esophagitis
Keywords: EoE; Eosinophil; Esophagitis
MeSH Terms: conditions — Eosinophilic Esophagitis; Esophagitis | interventions — AK002

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Subjects in this arm will receive 6 monthly doses of placebo.
  Interventions: Other: Placebo
- 1 mg/kg of lirentelimab (AK002) (Experimental): Subjects in this arm will receive 6 monthly doses of lirentelimab (AK002) (1mg/kg).
  Interventions: Drug: lirentelimab (AK002)
- 3 mg/kg of lirentelimab (AK002) (Experimental): Subjects in this arm will receive 6 monthly doses of lirentelimab (AK002): A first dose of 1 mg/kg, followed by 5 monthly doses of 3 mg/kg.
  Interventions: Drug: lirentelimab (AK002)

INTERVENTIONS:
Other: Placebo — Placebo
  Arms: Placebo
Drug: lirentelimab (AK002) — Lirentelimab (AK002) is a humanized non-fucosylated immunoglobulin G1 (IgG1) monoclonal antibody directed against Siglec-8.
  Arms: 1 mg/kg of lirentelimab (AK002); 3 mg/kg of lirentelimab (AK002)

SUMMARY:
This is a Phase 2/3, multi-center, randomized, double-blind, placebo-controlled study to assess the efficacy and safety of lirentelimab (AK002) given monthly for 6 doses in adult and adolescent patients with active eosinophilic esophagitis. Subjects who complete the randomized, double-blind, placebo-controlled treatment may have the option to receive 6 doses of open-label lirentelimab (AK002) through the OLE Period of the study.

ELIGIBILITY:
Key Inclusion Criteria:

1. Male or female aged ≥12 and ≤80 years at the time of signing ICF.
2. Confirmed diagnosis of EoE and esophageal intraepithelial eosinophilic infiltration of ≥15 eosinophils/hpf in 1 hpf from a biopsy collected during the Screening EGD without any other cause for the esophageal eosinophilia.
3. History (by patient report) of an average of ≥2 episodes of dysphagia with intake of solid foods per week during the 4 weeks prior to Screening.
4. Subjects must have failed or not be adequately controlled on standard of care treatments for EoE symptoms, which could include PPI, systemic or topical corticosteroids, and/or diet, among others.
5. If on an allowed treatment for EoE, stable dose for at least 4 weeks prior to Screening and willingness to continue that dose for the study duration.
6. If patient is on pre-existing dietary restrictions, willingness to maintain dietary restrictions throughout the study, as much as possible.
7. Able and willing to comply with all study procedures.
8. Female subjects must be either post-menopausal for at least 1 year with FSH level >30 mIU/mL at Screening or surgically sterile (tubal ligation,hysterectomy, or bilateral oophorectomy) for at least 3 months, or if of childbearing potential, have a negative pregnancy test and agree to use dual methods of contraception, or abstain from sexual activity from screening until the end of the study, or for 120 days following the last dose of study drug, whichever is longer. Male subjects with female partners of childbearing potential must agree to use a highly effective method of contraception from Screening until the end of the study or for 120 days following the last dose of study drug,whichever is longer. All fertile men with female partners of childbearing potential should be instructed to contact the Investigator immediately if they suspect their partner might be pregnant at any time during study participation.

Key Exclusion Criteria:

1. Concomitant EG, EoD, or eosinophilic colitis (EC).
2. EG and/or EoD (≥30 eosinophils/hpf in 5 hpf in the stomach and/or ≥30 eosinophils/hpf in 3 hpf in the duodenum) as determined by central histology assessment of biopsies collected during the Screening EGD.
3. Causes of esophageal eosinophilia other than EoE or one the following: hypereosinophilic syndrome, eosinophilic granulomatosis with polyangiitis, or peripheral blood absolute eosinophil count of >1500 eosinophils/μL.
4. History of inflammatory bowel disease, celiac disease, achalasia, and/or esophageal surgery.
5. Any esophageal stricture unable to be passed with a standard diagnostic 9 mm to 10 mm upper endoscope or any critical esophageal stricture that requires dilation during screening.
6. History of bleeding disorders or esophageal varices.
7. History of malignancy; except carcinoma in situ, early stage prostate cancer, or non-melanoma skin cancers. However, cancers that have been in remission for more than 5 years and are considered cured, can be enrolled (with the exception of breast cancer). All history of malignancy (including diagnosis, dates, and compliance with cancer screening recommendations) must be documented and certified by the Investigator, along with the statement that in their clinical judgment the tissue eosinophilia is attributable to EGID, rather than recurrence of malignancy.
8. Active Helicobacter pylori infection (as determined by central histology staining of the biopsy collected during the Screening EGD), unless treated and confirmed to be negative prior to randomization and symptoms remain consistent.
9. Positive Ova and Parasite (O&P) test at Screening, seropositive for Strongyloides stercoralis at Screening, and/or treatment for a clinically significant helminthic parasitic infection within 6 months of Screening.
10. Seropositive for HIV or hepatitis at Screening, except for vaccinated patients or patients with a history of hepatitis that has since resolved.
11. Prior exposure to AK002 or hypersensitivity to any constituent of AK002.
12. Change in dose of inhaled corticosteroids, nasal corticosteroids, PPI, and/or diet therapy within 4 weeks prior to Screening.
13. Use of oral corticosteroids (swallowed topical or systemic corticosteroids) within 8 weeks prior to Screening.
14. Use of any biologics or medications that may interfere with the study, such as immunosuppressive or immunomodulatory drugs including azathioprine, JAK inhibitors, 6-mercaptopurine, methotrexate, cyclosporine, tacrolimus, anti-TNF, anti-IL-4 receptor, e.g., dupilumab), anti-IL-5 (e.g., mepolizumab), anti-IL-5 receptor (e.g., benralizumab), anti-IL-13 (e.g., lebrikizumab), anti-IgE (e.g., omalizumab), within 12 weeks prior to Screening.
15. Participation in a concurrent interventional study with the last intervention occurring within 30 days prior to administration of study drug or 90 days or 5 half-lives, whichever is longer, for biologic products.
16. Vaccination with live attenuated vaccines ≤30 days prior to initiation of treatment in the study, during the treatment period, or vaccination expected ≤5 half-lives (≤4 months) following study drug administration.
17. Treatment with chemotherapy or radiotherapy in the preceding 6 months.
18. Presence of abnormal laboratory values considered by the Investigator to be clinically significant.
19. Any disease, condition (medical or surgical), or cardiac abnormality, which in the opinion of the Investigator, would place the subject at increased risk.
20. Known history of alcohol, drug, or other substance abuse or dependence.
21. Women who are pregnant, breastfeeding, or planning to become pregnant while participating in the study.
22. Any other reason that in the opinion of the Investigator or Medical Monitor makes the patient unsuitable for enrollment.

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 277 (Actual)
Dates: Start 2020-07-06 (Actual); Primary Completion 2021-06-04 (Actual); Study Completion 2022-01-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig Paterson, MD, Study Director — Allakos Inc.
Locations (70):
- United States (65):
  - Allakos Investigational Site, Birmingham, Alabama
  - Allakos Investigational Site, Huntsville, Alabama
  - Allakos Investigational Site, Gilbert, Arizona
  - Allakos Investigational Site, Phoenix, Arizona
  - Allakos Investigational Site, Scottsdale, Arizona
  - Allakos Investigational Site, Little Rock, Arkansas
  - Allakos Investigational Site, La Jolla, California
  - Allakos Investigational Site, Los Angeles, California
  - Allakos Investigational Site, Oakland, California
  - Allakos Investigational Site, Santa Monica, California
  - Allakos Investigational Site, Tustin, California
  - Allakos Investigational Site, Ventura, California
  - Allakos Investigational Site, Walnut Creek, California
  - Allakos Investigational Site, Aurora, Colorado
  - Allakos Investigational Site, Centennial, Colorado
  - Allakos Investigational Site, Brandon, Florida
  - Allakos Investigational Site, Edgewater, Florida
  - Allakos Investigational Site, Jacksonville, Florida
  - Allakos Investigational Site, Miami, Florida
  - Allakos Investigational Site, Orlando, Florida
  - Allakos Investigational Site, Tampa, Florida
  - Allakos Investigational Site, Atlanta, Georgia
  - Allakos Investigational Site, Columbus, Georgia
  - Allakos Investigational Site, Chicago, Illinois
  - Allakos Investigational Site, Indianapolis, Indiana
  - Allakos Investigational Site, Iowa City, Iowa
  - Allakos Investigational Site, Lexington, Kentucky
  - Allakos Investigational Site, Crowley, Louisiana
  - Allakos Investigational Site, Chevy Chase, Maryland
  - Allakos Investigational Site, Boston, Massachusetts
  - Allakos Investigational Site, Ann Arbor, Michigan
  - Allakos Investigational Site, Troy, Michigan
  - Allakos Investigational Site, Kansas City, Missouri
  - Allakos Investigational Site, Kalispell, Montana
  - Allakos Investigational Site, Las Vegas, Nevada
  - Allakos Investigational Site, Reno, Nevada
  - Allakos Investigational Site, Great Neck, New York
  - Allakos Investigational Site, New York, New York
  - Allakos Investigational Site, Asheville, North Carolina
  - Allakos Investigational Site, Chapel Hill, North Carolina
  - Allakos Investigational Site, Charlotte, North Carolina
  - Allakos Investigational Site, Durham, North Carolina
  - Allakos Investigational Site, High Point, North Carolina
  - Allakos Investigational Site, Rocky Mount, North Carolina
  - Allakos Investigational Site, Akron, Ohio
  - Allakos Investigational Site, Cincinnati, Ohio
  - Allakos Investigational Site, Cleveland, Ohio
  - Allakos Investigational Site, Dayton, Ohio
  - Allakos Investigational Site, Mentor, Ohio
  - Allakos Investigational Site, Oklahoma City, Oklahoma
  - Allakos Investigational Site, Danville, Pennsylvania
  - Allakos Investigational Site, Philadelphia, Pennsylvania
  - Allakos Investigational Site, Greenville, South Carolina
  - Allakos Investigational Site, Chattanooga, Tennessee
  - Allakos Investigational Site, Hixson, Tennessee
  - Allakos Investigational Site, Nashville, Tennessee
  - Allakos Investigational Site, Austin, Texas
  - Allakos Investigational Site, Garland, Texas
  - Allakos Investigational Site, San Antonio, Texas
  - Allakos Investigational Site, Ogden, Utah
  - Allakos Investigational Site, Riverton, Utah
  - Allakos Investigational Site, Salt Lake City, Utah
  - Allakos Investigational Site, Sandy City, Utah
  - Allakos Investigational Site, Leesburg, Virginia
  - Allakos Investigational Site, Seattle, Washington
- Australia (4):
  - Allakos Investigational Site, Adelaide, South Australia
  - Allakos Investigational Site, Elizabeth Vale, South Australia
  - Allakos Investigational Site, Box Hill, Victoria
  - Allakos Investigational Site, Prahran, Victoria
- Allakos Investigational Site, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | 1 mg/kg of Lirentelimab (AK002) | 3 mg/kg of Lirentelimab (AK002)
Started | 92 | 93 | 91
Completed | 89 | 89 | 85
Not Completed | 3 | 4 | 6

BASELINE CHARACTERISTICS:
Population: Modified Intention-to-treat
Groups:
- AK002 1 mg/kg: Patients randomized to 1, 1, 1, 1, 1, 1 mg/kg on Days 1, 29, 57, 85, 113, 141
- AK002 3 mg/kg: Patients randomized to 1, 3, 3, 3, 3, 3 mg/kg on Days 1, 29, 57, 85, 113, 141
- Placebo: Patients randomized to placebo on Days, 1, 29, 57, 85, 113, 141
- Total: Total of all reporting groups
Arm/Group | AK002 1 mg/kg | AK002 3 mg/kg | Placebo | Total
Number analyzed (Participants) | 93 | 91 | 92 | 276
Age, Continuous [Median (Full Range); unit: years] | 34 [12 to 67] | 29 [12 to 69] | 32 [12 to 70] | 32 [12 to 70]
Age, Customized [Count of Participants; unit: Participants]
  <18 years | 17 | 17 | 17 | 51
  >=18 years | 76 | 74 | 75 | 225
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 26 | 37 | 103
  Male | 53 | 65 | 55 | 173
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 5 | 9 | 22
  Not Hispanic or Latino | 84 | 82 | 82 | 248
  Unknown or Not Reported | 1 | 4 | 1 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 1 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 2 | 2 | 5 | 9
  White | 87 | 85 | 84 | 256
  More than one race | 2 | 0 | 1 | 3
  Unknown or Not Reported | 1 | 2 | 1 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 91 | 88 | 88 | 267
  Netherlands | 1 | 1 | 1 | 3
  Australia | 1 | 2 | 3 | 6
Baseline Esophageal Eosinophil Count [Mean (Standard Deviation); unit: Eosinophils/HPF] — Number of eosinophils per high power field (HPF) in esophageal mucosa
  Eosinophils/HPF | 61.2 (35.3) | 58.9 (32.8) | 58.8 (32.8) | 59.7 (33.6)
Dysphagia Symptom Questionnaire (DSQ) Total Score [Mean (Standard Deviation); unit: Score on a scale] — The DSQ is used to measure the frequency and intensity of dysphagia. DSQ scores can range from 0 to 84, with a lower score indicating less frequent or less severe dysphagia.
  Score on a scale | 36.4 (12.0) | 34.2 (11.8) | 35.2 (12.1) | 35.3 (11.9)

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects Who Achieve a Peak Esophageal Intraepithelial Count of ≤6 Eosinophils/Hpf at Week 24
Description: Esophageal intraepithelial eosinophil count obtained by esophageal endoscopy with biopsies.
Time Frame: At Week 24
Population: Modified Intention-to-treat
Measure: Count of Participants; unit: Participants
Arm/Group | 1 mg/kg of Lirentelimab (AK002) | 3 mg/kg of Lirentelimab (AK002) | Placebo
Number analyzed (Participants) | 93 | 91 | 92
Participants | 86 | 80 | 10
Statistical Analysis 1: Comparison: 1 mg/kg of Lirentelimab (AK002) vs Placebo; Test type: Superiority; p < 0.0001, Fisher Exact; Percent Difference from Placebo = 81.6, 95% CI 2-sided [71.5 to 89.0]
Statistical Analysis 2: Comparison: 3 mg/kg of Lirentelimab (AK002) vs Placebo; Test type: Superiority; p < 0.0001, Fisher Exact; Percent Difference from Placebo = 77.0, 95% CI 2-sided [66.1 to 85.4]

2. Primary Outcome: Change in Dysphagia Symptom Questionnaire (DSQ) Score From Baseline to Weeks 23-24.
Description: The DSQ is used to measure the frequency and intensity of dysphagia. DSQ scores can range from 0 to 84, with a lower score indicating less-frequent or less-severe dysphagia.
Time Frame: Baseline to Weeks 23-24
Population: Modified Intention-to-treat
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | 1 mg/kg of Lirentelimab (AK002) | 3 mg/kg of Lirentelimab (AK002) | Placebo
Number analyzed (Participants) | 93 | 91 | 92
Score on a scale | -11.9 (1.8) | -17.4 (1.8) | -14.6 (1.8)
Statistical Analysis 1: Comparison: 1 mg/kg of Lirentelimab (AK002) vs Placebo; Test type: Superiority; p = 0.2470, ANCOVA; LSM Difference from Placebo = 2.7, 95% CI 2-sided [-1.9 to 7.3]
Statistical Analysis 2: Comparison: 3 mg/kg of Lirentelimab (AK002) vs Placebo; Test type: Superiority; p = 0.2372, ANCOVA; LSM Difference from Placebo = -2.8, 95% CI 2-sided [-7.3 to 1.8]

3. Secondary Outcome: Percent Change in Peak Esophageal Intraepithelial Eosinophil Count From Baseline to Week 24
Description: Esophageal intraepithelial eosinophil count obtained by esophageal endoscopy with biopsies. A greater esophageal intraepithelial eosinophil count from baseline indicates worsening disease.
Time Frame: Baseline to Week 24
Population: Modified Intention-to-treat
Measure: Mean (Standard Deviation); unit: Percentage of Change
Arm/Group | 1 mg/kg of Lirentelimab (AK002) | 3 mg/kg of Lirentelimab (AK002) | Placebo
Number analyzed (Participants) | 93 | 91 | 92
Percentage of Change | -98.9 (5.6) | -99.6 (1.0) | -3.1 (76.0)
Statistical Analysis 1: Comparison: 1 mg/kg of Lirentelimab (AK002) vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA; LSM Difference from Placebo = -95.7, 95% CI 2-sided [-109 to -82.4]
Statistical Analysis 2: Comparison: 3 mg/kg of Lirentelimab (AK002) vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA; LSM Difference from Placebo = -96.2, 95% CI 2-sided [-110 to -82.5]

4. Secondary Outcome: Subjects Achieving Peak Esophageal Intraepithelial Eosinophil Count of ≤1 Eosinophil/Hpf at Week 24
Description: Esophageal intraepithelial eosinophil count obtained by esophageal endoscopy with biopsies.
Time Frame: At Week 24
Population: Modified Intention-to-treat
Measure: Count of Participants; unit: Participants
Arm/Group | 1 mg/kg of Lirentelimab (AK002) | 3 mg/kg of Lirentelimab (AK002) | Placebo
Number analyzed (Participants) | 93 | 91 | 92
Participants | 82 | 77 | 4
Statistical Analysis 1: Comparison: 1 mg/kg of Lirentelimab (AK002) vs Placebo; Test type: Superiority; p < 0.0001, Fisher Exact; Percent Difference from Placebo = 83.8, 95% CI 2-sided [74.4 to 90.8]
Statistical Analysis 2: Comparison: 3 mg/kg of Lirentelimab (AK002) vs Placebo; Test type: Superiority; p < 0.0001, Fisher Exact; Percent Difference from Placebo = 80.3, 95% CI 2-sided [69.8 to 87.9]

5. Secondary Outcome: Subjects Achieving Peak Esophageal Intraepithelial Eosinophil Count of <15 Eosinophils/Hpf at Week 24
Description: Esophageal intraepithelial eosinophil count obtained by esophageal endoscopy with biopsies.
Time Frame: At Week 24
Population: Modified Intention-to-treat
Measure: Count of Participants; unit: Participants
Arm/Group | 1 mg/kg of Lirentelimab (AK002) | 3 mg/kg of Lirentelimab (AK002) | Placebo
Number analyzed (Participants) | 93 | 91 | 92
Participants | 86 | 80 | 14
Statistical Analysis 1: Comparison: 1 mg/kg of Lirentelimab (AK002) vs Placebo; Test type: Superiority; p < 0.0001, Fisher Exact; Percent Difference from Placebo = 77.3, 95% CI 2-sided [66.4 to 85.5]
Statistical Analysis 2: Comparison: 3 mg/kg of Lirentelimab (AK002) vs Placebo; Test type: Superiority; p < 0.0001, Fisher Exact; Percent Difference from Placebo = 72.7, 95% CI 2-sided [61.3 to 81.9]

6. Secondary Outcome: Number of Treatment Responders
Description: Treatment responders defined by >30% improvement in symptoms (DSQ) at Weeks 23-24 and peak intraepithelial eosinophilic count of ≤6 cells/hpf at Week 24
Time Frame: At Weeks 23-24 and Week 24, Respectively
Population: Modified Intention-to-treat
Measure: Count of Participants; unit: Participants
Arm/Group | 1 mg/kg of Lirentelimab (AK002) | 3 mg/kg of Lirentelimab (AK002) | Placebo
Number analyzed (Participants) | 93 | 91 | 92
Participants | 42 | 53 | 8
Statistical Analysis 1: Comparison: 1 mg/kg of Lirentelimab (AK002) vs Placebo; Test type: Superiority; p < 0.0001, Fisher Exact; Percent Difference from Placebo = 36.5, 95% CI 2-sided [22.9 to 49.5]
Statistical Analysis 2: Comparison: 3 mg/kg of Lirentelimab (AK002) vs Placebo; Test type: Superiority; p < 0.0001, Fisher Exact; Percent Difference from Placebo = 49.5, 95% CI 2-sided [35.9 to 61.0]

7. Secondary Outcome: Subjects Who Achieve >50% Reduction in DSQ Score From Baseline to Weeks 23-24
Description: as for outcome 2
Time Frame: Weeks 23-24
Population: Modified Intention-to-treat
Measure: Count of Participants; unit: Participants
Arm/Group | 1 mg/kg of Lirentelimab (AK002) | 3 mg/kg of Lirentelimab (AK002) | Placebo
Number analyzed (Participants) | 93 | 91 | 92
Participants | 40 | 48 | 44
Statistical Analysis 1: Comparison: 1 mg/kg of Lirentelimab (AK002) vs Placebo; Test type: Superiority; p = 0.5561, Fisher Exact; Percent Difference from Placebo = -4.8, 95% CI 2-sided [-19.2 to 10.0]
Statistical Analysis 2: Comparison: 3 mg/kg of Lirentelimab (AK002) vs Placebo; Test type: Superiority; p = 0.5554, Fisher Exact; Percent Difference from Placebo = 4.9, 95% CI 2-sided [-9.9 to 19.6]

8. Secondary Outcome: Percent Change in DSQ Score From Baseline to Weeks 23-24
Description: as for outcome 2
Time Frame: Baseline to Weeks 23-24
Population: Modified Intention-to-treat
Measure: Mean (Standard Deviation); unit: Percentage of Change
Arm/Group | 1 mg/kg of Lirentelimab (AK002) | 3 mg/kg of Lirentelimab (AK002) | Placebo
Number analyzed (Participants) | 93 | 91 | 92
Percentage of Change | -36.3 (51.4) | -56.2 (39.8) | -36.2 (82.5)
Statistical Analysis 1: Comparison: 1 mg/kg of Lirentelimab (AK002) vs Placebo; Test type: Superiority; p = 0.9506, ANCOVA; LSM Difference from Placebo = -0.6, 95% CI 2-sided [-18.1 to 17.0]
Statistical Analysis 2: Comparison: 3 mg/kg of Lirentelimab (AK002) vs Placebo; Test type: Superiority; p = 0.0511, ANCOVA; LSM Difference from Placebo = -17.6, 95% CI 2-sided [-35.4 to 0.1]

9. Secondary Outcome: Change in Biweekly Mean DSQ Over Time Using MMRM
Description: as for outcome 2
Time Frame: Baseline to Weeks 23-24
Population: Modified Intention-to-treat
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | 1 mg/kg of Lirentelimab (AK002) | 3 mg/kg of Lirentelimab (AK002) | Placebo
Number analyzed (Participants) | 93 | 91 | 92
Score on a Scale
  Weeks 1-2 | -4.2 (9.0) | -6.5 (9.9) | -6.2 (10.1)
  Weeks 3-4 | -7.2 (10.9) | -8.4 (12.4) | -8.1 (11.3)
  Weeks 5-6 | -8.4 (12.9) | -11.5 (14.1) | -11.7 (12.0)
  Weeks 7-8 | -10 (13.6) | -12.2 (13.8) | -12.0 (14.5)
  Weeks 9-10 | -10.5 (14.5) | -14.7 (14.7) | -13.6 (13.4)
  Weeks 11-12 | -11.1 (14.4) | -15.0 (14.0) | -13.3 (14.7)
  Weeks 13-14 | -11.7 (15.0) | -16.5 (14.6) | -15.0 (14.4)
  Weeks 15-16 | -11.4 (15.8) | -17.0 (14.8) | -13.5 (15.6)
  Weeks 17-18 | -12.4 (15.6) | -17.5 (14.4) | -14.4 (15.8)
  Weeks 19-20 | -12.1 (15.6) | -17.8 (14.5) | -14.8 (17.0)
  Weeks 21-22 | -12.4 (14.7) | -17.6 (15.0) | -15.7 (17.1)
  Weeks 23-24 | -12.1 (15.0) | -18.0 (14.7) | -14.6 (17.5)
Statistical Analysis 1: Comparison: 1 mg/kg of Lirentelimab (AK002) vs Placebo; Weeks 23-24 Change from Baseline; Test type: Superiority; p = 0.2007, Mixed Models Analysis; LSM Difference from Placebo = 2.6, 95% CI 2-sided [-1.4 to 6.7]
Statistical Analysis 2: Comparison: 3 mg/kg of Lirentelimab (AK002) vs Placebo; Weeks 23-24 Change from Baseline; Test type: Superiority; p = 0.1889, Mixed Models Analysis; LSM Difference from Placebo = -2.7, 95% CI 2-sided [-6.8 to 1.3]

10. Secondary Outcome: Change in EoE Reference Score for Endoscopic Abnormalities (EREFS) From Baseline to Week 24
Description: EoE esophageal characteristics analyzed based on the EoE-EREFS, a scoring system for inflammatory and remodeling features of disease. The overall total score ranges from 0 to 18 with higher number indicating worse disease.
Time Frame: Baseline to Week 24
Population: Modified Intention-to-treat
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | 1 mg/kg of Lirentelimab (AK002) | 3 mg/kg of Lirentelimab (AK002) | Placebo
Number analyzed (Participants) | 93 | 91 | 92
Score on a scale | -1.3 (3.2) | -1.0 (3.9) | -1.5 (3.8)
Statistical Analysis 1: Comparison: 1 mg/kg of Lirentelimab (AK002) vs Placebo; Test type: Superiority; p = 0.4980, ANCOVA; LSM Difference from Placebo = -0.3, 95% CI 2-sided [-1.3 to 0.6]
Statistical Analysis 2: Comparison: 3 mg/kg of Lirentelimab (AK002) vs Placebo; Test type: Superiority; p = 0.6390, ANCOVA; LSM Difference from Placebo = 0.2, 95% CI 2-sided [-0.7 to 1.2]

ADVERSE EVENTS:
Time Frame: Baseline up to Day 197
Arm/Group | 1 mg/kg of Lirentelimab (AK002) | 3 mg/kg of Lirentelimab (AK002) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/93 | 0/91 | 0/92
Serious Adverse Events (participants affected / at risk) | 4/93 | 3/91 | 2/92
Other Adverse Events (participants affected / at risk) | 37/93 | 39/91 | 23/92
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 1 mg/kg of Lirentelimab (AK002) (N=93) | 3 mg/kg of Lirentelimab (AK002) (N=91) | Placebo (N=92)
Palpitations (Cardiac disorders) | 1 | 0 | 0
Eye swelling (Eye disorders) | 0 | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0
Angioedema (Immune system disorders) | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 2 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Lip swelling (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Epistaxis (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 mg/kg of Lirentelimab (AK002) (N=93) | 3 mg/kg of Lirentelimab (AK002) (N=91) | Placebo (N=92)
Nausea (Gastrointestinal disorders) | 4 (4) | 4 (6) | 8 (12)
Vomiting (Gastrointestinal disorders) | 1 (1) | 5 (6) | 7 (8)
Fatigue (General disorders) | 3 (7) | 3 (3) | 5 (6)
Infusion related reaction (Injury, poisoning and procedural complications) | 24 (36) | 33 (41) | 11 (27)
Blood creatine phosphokinase increased (Investigations) | 6 (6) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 8 (17) | 7 (12) | 6 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Clinical Trial Agreement contains a limit on publication of results following completion of the trial. PIs are not allowed to publish results until a joint publication for the multicenter study or a set period of time. After that time, PIs may only publish results from their portion of the study.

DOCUMENTS (2):
  • Study Protocol (2021-11-05): https://cdn.clinicaltrials.gov/large-docs/08/NCT04322708/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-10): https://cdn.clinicaltrials.gov/large-docs/08/NCT04322708/SAP_001.pdf